CLINICAL TRIAL: NCT03372954
Title: Retrograde Application of Bone Marrow Aspirate Concentrate (BMAC) Through Coronary Sinus in Patients With Congestive Heart Failure of Ischemic Etiology
Brief Title: Retrograde Application of Bone Marrow Aspirate Concentrate
Acronym: Retro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-Retro
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone marrow autologous cells concentrate (BMAC) (Experimental): retrograde administration on non-selected BMAC via coronary sinus
  Interventions: Drug: BMAC
- Control (Placebo Comparator): standard treatment o heart failure
  Interventions: Drug: BMAC

INTERVENTIONS:
Drug: BMAC — retrograde administration on non-selected BMAC via coronary sinus

SUMMARY:
The aim of our prospective randomised study is to assess the efficacy of the retrograde application of non-selected bone marrow autologous cells concentrate (BMAC) in patients with heart failure with reduced ejection fraction of left ventricle (HFREF) of ischemic aetiology. The evaluated preparation is concentrated BMAC, obtained using Harvest SmartPReP2 technology.

DETAILED DESCRIPTION:
Our assumption is that non-selected BMAC administrations will lead to improvements in the left ventricular ejection fraction (LV EF), the left ventricular end-systolic and end-diastolic diameters and volumes (measured with magnetic resonance imaging) compared to standard heart failure therapy.

Furthermore, it will be associated with improved exercise tolerance in the six-minute corridor walk test and an improvement in the life quality of patients without increasing the incidence of severe ventricular arrythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure and left ventricular ejection fraction ≤ 40% with coronary artery disease and with symptoms of heart failure in the NYHA class ≥ 3 on standard heart failure therapy for 3 months and in a stabilised state for at least 1 month
* Age ≥18 years
* Informed, written consent by the patient
* Ability to comply fully with the study protocol
* Negative pregnancy test (and effective contraception) in women with childbearing potential

Exclusion Criteria:

* Previous bone marrow disease (especially myelodysplastic syndrome or non-Hodgkin's lymphoma)
* Acute myocardial infarction ˂ 1 week
* Active infection or antibiotics treatment ˂ 1 week
* Previous malingant ventricular arrhythmias without cardioverter-defibrilator (ICD) implantation
* Anemia (HTC≤28%), leukocythosis (≥ 14.000/mm3) or thrombocytopenia (≤50.000/mm3)
* Previous bleeding diathesis
* Need for hematopoietic growth factor treatment (e.g. erythropoetin, G-CSF)
* Impossibility of aspiration 240ml of bone marrow
* Hepathopathy or cirrhosis (bilirubin, ALT or AST ≥ 2,5x upper limit of normal)
* Terminal renal insufficiency or haemodyalysis
* Uncontrolled hypertension
* Need for high dose (> 7.5mg/day) corticotherapy within the next 6 months
* Inability to stop anticoagulation therapy (>72 hours) before bone marrow aspiration
* Known malignancies requiring actino or chemotherapy, or previous actinotherapy
* Patients with a BMI >40
* Known allergy to contrast agents
* Other comorbidities with a life expectancy of 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular end-systolic diameter (LVESd) | 12 month
  Left ventricular end-systolic diameter
Left ventricular end-systolic volume (LVESV) | 12 month
  Left ventricular end-systolic volume
Left ventricular end-diastolic diameter (LVEDd) | 12 month
  Left ventricular end-diastolic diameter
Left ventricular end-diastolic volume (LVEDV) | 12 month
  Left ventricular end-diastolic volume
ejection fraction of left ventricle (EF LV) | 12 month
  ejection fraction of left ventricle

SECONDARY OUTCOMES:
corridor walk test | 12 month
  walk distance in 6 min corridor walk test
QoL | 12 month
  Quality of patients´ life using the Minnesota questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Leoš Pleva, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There exists no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Derived] Pleva L, Kukla P, Vitkova K, Prochazka V. Rationale and design of a prospective, randomised study of retrograde application of bone marrow aspirate concentrate (BMAC) through coronary sinus in patients with congestive heart failure of ischemic etiology (the RETRO study). BMC Cardiovasc Disord. 2019 Jan 31;19(1):32. doi: 10.1186/s12872-019-1011-9. PMID 30704414